CLINICAL TRIAL: NCT04307953
Title: Saracatinib Trial TO Prevent FOP
Acronym: STOPFOP
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: Royal National Orthopaedic Hospital NHS Trust (Other); Klinikum Garmisch-Patenkirchen (Other); University of Oxford (Other); Brigham and Women's Hospital (Other); AstraZeneca (Industry); Innovative Medicines Initiative (Other)
Responsible Party: Principal Investigator, Elisabeth MW Eekhoff, Coordinating Principal Investigator, Amsterdam UMC, location VUmc
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STOPFOP1; 2019-003324-20 (EudraCT Number); NL71401.029.19 (Other: Dutch Competent Authority)
Record Dates: First submitted 2020-03-11; First posted 2020-03-13 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-04

CONDITIONS: Fibrodysplasia Ossificans Progressiva
Keywords: Fibrodysplasia Ossificans Progressiva; AZD0530; Saracatinib; Stone man syndrome; FOP
MeSH Terms: conditions — Myositis Ossificans | interventions — saracatinib

STUDY DESIGN:
Intervention Model Description: 6-month double blind randomized controlled trial of AZD0530 versus placebo, followed by a 12 month open label extension phase
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AZD0530 (Experimental)
  Interventions: Drug: AZD0530 Difumarate
- Placebo/AZD0530 (Experimental)
  Interventions: Drug: Matching placebo

INTERVENTIONS:
Drug: AZD0530 Difumarate — AZD0530 for the duration of the trial
  Other Names: Saracatinib
  Arms: AZD0530
Drug: Matching placebo — Matching placebo during 6 month RCT, AZD0530 thereafter
  Arms: Placebo/AZD0530

SUMMARY:
This is a phase 2 study, designed as a European multicentre 6-month double blind random-ized controlled trial (RCT) of AZD0530 versus matched placebo, followed by a 12 month trial comparing open-label extended AZD0530 treatment with historical control data.

Study population: Male and female adult patients aged 18 years and older with a diagnosis of FOP who meet the inclusion (active disease) and exclusion criteria will be eligible for participation in this study. The total number of enrolled patients will be 20.

Intervention: Patients will be randomized to receive either AZD0530 100mg once daily or matched placebo, taken orally for the first 6 months, immediately followed by an open-label extension in which all patients will receive AZD0530 100mg once daily oral dose for a further 12 months.

Endpoints: Endpoints include objective change in heterotopic bone volume measured by low-dose whole-body computer tomography (CT) , [18F] NaF Positron Emission Tomography (PET) activity and patient reported outcome measures.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 18-65 with a clinical diagnosis of FOP at screening, including congenital malformation of the great toes and a history of spontaneous or injury-induced heterotopic ossification (HO), and have a confirmed classic FOP phenotype by the documentation of an ACVR1R206H/+ or variant genomic sequence.

   1. Female participants who are women of child-bearing potential will be required to use a highly effective method of contraception as defined in section 5.4, in combination with a condom or diaphragm or cervical/vault caps with spermicidal foam/gel/film/suppository), from the time of enrolment until 4 weeks after final dose of study drug, unless practicing true sexual abstinence as defined in section 5.4.
   2. Male participants will be required to avoid procreative sexual intercourse with women of child-bearing potential from time of enrollment until 4 weeks after final dose of study drug through use of highly effective contraceptive methods. Male participants with a pregnant female partner will be required to use a condom for the duration of the study and for 4 weeks final dose of study drug. Male study participants will not be permitted to donate sperm for from the time of enrolment and until 4 weeks after final dose of study drug.
2. Participants will have to be able to understand and complete study and willing to sign informed consent (IC). They have to be able to attend and comply with the study visits and related activities, adhere to all study-related restrictions, and able to undergo procedures such as PET and CT imaging.

Exclusion Criteria:

1. Not willing to strictly adhere to the reproductive restrictions as defined in section 5.4
2. Women who are pregnant or breast-feeding (from the time 3 months prior to 4 weeks after completion of participation in the study)
3. The presence of significant concomitant illness or history of significant illness such as cardiac, respiratory, renal, rheumatologic, neurologic, psychiatric, endocrine, metabolic, lymphatic disease, or infectious disease, that might confound the results of the study or pose additional risk to the patient;
4. Evidence of active bleeding (including hematuria or hematochezia,) acute or chronic gastrointestinal illness, inflammatory bowel disease, or mucositis
5. Malignant disease / cancer requiring treatment in the past 3 years (except some primary non melanoma skin cancer);
6. Severely impaired renal function defined as estimated glomerular filtration rate <30 mL/min/1.73 m2 calculated by the Modification of Diet in Renal Disease equation;
7. Showing uncontrolled diabetes mellitus with an HbA1C > 9%;
8. Significant viral illness or active infections at screening or randomisation; Subjects should not have subacute or acute fevers of >101 degrees F at time of screening or randomisation
9. Evidence of prolonged QT interval at screening or randomization (defined as QTc of >450 ms) .or known congenital long-QT syndrome.
10. Neutropenia defined as an absolute neutrophil count of <1,500/µl,
11. Thrombocytopenia defined as platelet count <100 × 103/µl,
12. Current blood clotting or bleeding disorder, or significantly abnormal INR-prothrombin time or partial thromboplastin time at screening, or clinically significant abnormalities in other screening laboratories, including significant abnormalities in vitamin B12 or thyroid function tests would be cause for exclusion.-
13. Abnormal liver function test results defined as aspartate aminotransferase (AST) >2.0 x upper limit of normal (ULN); alanine aminotransferase (ALT) >2.0 x ULN; and / or total bilirubin >1.5 x ULN;
14. Known allergy or intolerance to AZD0530 or any excipients used in the investigational medicinal products.
15. Simultaneous participation in another interventional clinical study or a non-interventional study with imaging measures or invasive procedures (eg. collection of blood or tissue samples); Participation in the FOP Connection Registry (www.fopconnection.org) or other studies in which patients completed study questionnaires are possible.
16. Treatment with another investigational or drug that might interfere with HO formation and the interpretation of the study drug in the last 90 days
17. Current use or history of regular alcohol consumption exceeding 14 units/week (6 glasses of 13.0% wine (175ml), 6 pints of 4.0% lager or ale (568ml), 5 pints of 4.5% cider (568 ml) or 14 glasses of 10.0% spirits (25ml)) within 6 months of screening.
18. Currently active metabolic bone disease, other than FOP.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-08-05 (Actual); Primary Completion 2025-05-06 (Estimated); Study Completion 2025-05-06 (Estimated)

PRIMARY OUTCOMES:
The objective change between the two arms measured in heterotopic bone volume measured by low-dose whole body CT over the initial 6 month RCT | Baseline, month 6

SECONDARY OUTCOMES:
Safety and tolerability assessments are the incidence and severity of adverse events (AE) during the RCT at the end of week 28. | Baseline, month 6 (+overall duration study)
The change in heterotopic bone volume measured by low-dose whole body CT over six-months treatment during open-label extension of AZD0530 compared to the previous placebo arm of the RCT | Baseline, month 6, month 12
The change in heterotopic bone volume measured by low-dose whole body CT over twelve-months treatment during open-label extension of AZD0530 compared to the historical data of Clementia (NCT02322255) | Baseline, month 6, month 12, month 18
Change in the volume of individual HO lesions | Baseline, month 6, month 12, month 18
  measured by low-dose whole body CT over the initial 6 month RCT and the change over twelve-months therapy during open-label extension of AZD0530 compared to the historical data of Clementia and compared to the 6 months placebo-arm.
Change in number of HO lesions measured by CT over the initial 6 month RCT and in addition the change over twelve-months during open-label extension of AZD0530 compared to the historical data of Clementia and compared to the 6 months placebo-arm. | Baseline, month 6, month 12, month 18
In patients with at least 1 active lesion at baseline: Change (and Area Under the Curve (AUC) analysis) of lesion activity | Baseline, month 6, month 12
  by 18F-NaF PET over the initial 6 month RCT and over months 6-12 compared to the 6 months RCT of the placebo arm, including change from baseline in 18F-NaF Standard Uptake Volume (SUVmean or peak) of individual active HO site
In patients with at least 1 active lesion at baseline: Change in number of active lesion on 18F-NaF PET from baseline to 6 and 12months | Baseline, month 6, month 12
Change and percent change from baseline in biomarkers of bone formation levels in serum over time. | Baseline, week 3 through month 18
  Including Total Procollagen Type 1 N-Terminal Propeptide (P1NP), Alkaline Phosphatase (AP) fasting cross-linked C-terminal telopeptide of type I colla-gen (βCTX). Selected genetic markers for FOP activity
Joint function assessment by physician at baseline and week 3, month 3,6,9,12,and18 by the cumulative analog joint involvement scale (CAJIS) and the quantitative detailed multi-joint assessment at baseline and month 6, 12 and 18 | baseline, week 3, month 3,6,9,12,and 18
Patient-reported global health status the 36-item Short Form Health Survey (SF-36) at baseline and week 3, month 3,6,9,12,and 18 | baseline, week 3, month 3,6,9,12,and 18
FOP disease activity assessed by movement disabilities and quality of life using FOP Independent Activity of Daily Living (FOP I-ADL) | baseline, week 3, month 3,6,9,12,and 18
Number of reported flare-ups by the patient | Each day (day 0-month18)
Pharmacokinetic measurements: blood for determination of plasma concentrations of AZD0530 (pre-dose)on the day of the study visits at 6, 12 and 18months | 6,12 and 18months

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth MW Eekhoff, MD, PhD, Principal Investigator — Amsterdam University Medical Center
Locations (3):
- Klinikum Garmish-Partenkirchen, Garmisch-Partenkirchen, Germany
- Amsterdam University Medical Center, Amsterdam, Netherlands
- Royal National Orthopaedic Hospital, London, United Kingdom

REFERENCES:
- [Derived] Smilde BJ, Stockklausner C, Keen R, Whittaker A, Bullock AN, von Delft A, van Schoor NM, Yu PB, Eekhoff EMW. Protocol paper: a multi-center, double-blinded, randomized, 6-month, placebo-controlled study followed by 12-month open label extension to evaluate the safety and efficacy of Saracatinib in Fibrodysplasia Ossificans Progressiva (STOPFOP). BMC Musculoskelet Disord. 2022 Jun 1;23(1):519. doi: 10.1186/s12891-022-05471-x. PMID 35650602